CLINICAL TRIAL: NCT02713477
Title: A Randomized, Open Label, Placebo-controlled, 4-sequence, 4-period, 4-treatment Crossover Study to Investigate the Postprandial Glucodynamic Response to Single Dose of Insulin Glargine/Lixisenatide Fixed Ratio Combination in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Postprandial Glucodynamic Response to Insulin Glargine/Lixisenatide Fixed Ratio Combination in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDY14115; U1111-1176-6235 (Other: UTN)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2016-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Insulin glargine/ lixisenatide dose 1 Test 1 (Experimental): Test 1 will be administered thru subcutaneous (SC) injection into one peri-umbilical site of the abdomen 1 hour prior to breakfast under fasted condition
  Interventions: Drug: Insulin glargine/ lixisenatide fixed-ratio combination HOE901/AVE0010
- Insulin glargine/ lixisenatide dose 2 Test 2 (Experimental): Test 2 will be administered thru SC injection into one peri-umbilical site of the abdomen 1 hour prior to breakfast under fasted condition
  Interventions: Drug: Insulin glargine/ lixisenatide fixed-ratio combination HOE901/AVE0010
- Placebo - Reference 1 (Placebo Comparator): Reference 1 will be administered thru SC injection into one peri-umbilical site of the abdomen 1 hour prior to breakfast under fasted condition
  Interventions: Drug: Placebo
- Insulin glargine (Lantus) - Reference 2 (Other): Reference 2 will be administered thru SC injection into one peri-umbilical site of the abdomen 1 hour pior to breakfast under fasted condition
  Interventions: Drug: Insulin glargine HOE901

INTERVENTIONS:
Drug: Insulin glargine/ lixisenatide fixed-ratio combination HOE901/AVE0010 — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Insulin glargine/ lixisenatide dose 1 Test 1; Insulin glargine/ lixisenatide dose 2 Test 2
Drug: Insulin glargine HOE901 — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Lantus
  Arms: Insulin glargine (Lantus) - Reference 2
Drug: Placebo — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Placebo - Reference 1

SUMMARY:
Primary Objective:

To assess the postprandial glucodynamic response to 2 doses of insulin glargine/lixisenatide fixed-ratio combination compared to placebo in Japanese patients with type 2 diabetes mellitus (T2DM).

Secondary Objectives:

* To assess the pharmacokinetics (PK) of lixisenatide following administration of 2 different doses of insulin glargine/lixisenatide fixed-ratio combination in Japanese patients with T2DM.
* To assess the postprandial glucodynamic response to insulin glargine/lixisenatide fixed-ratio combination compared to insulin glargine alone in Japanese patients with T2DM.
* To assess the safety and tolerability of insulin glargine/lixisenatide fixed-ratio combination in Japanese patients with T2DM.

DETAILED DESCRIPTION:
The total study duration per patient will be approximately 6 to 13 weeks that will consist of a 2-28 days of screening period, a 3-day treatment period, a 7-14 days of washout period, and 1-day end of study visit.

ELIGIBILITY:
Inclusion criteria :

* Japanese male or female patients with T2DM diagnosed for at least 1 year prior to the time of screening as established in the medical history.
* Patients aged 20 to 75 years at screening.
* Body mass index ≤35 kg/m^2 at screening.
* Glycohemoglobin ≥7.0% and ≤10.0% at screening.
* Fasting C-peptide ≥0.6 ng/mL at screening.

Exclusion criteria:

* Diabetes other than T2DM.
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening.
* History of hypoglycemia unawareness.
* Hemoglobinopathy or hemolytic anemia.
* History of myocardial infarction, stroke, or heart failure, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease.
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment.
* Personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (e.g., multiple endocrine neoplasia syndromes).
* If female, pregnancy or breast-feeding.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measurement of plasma glucose concentrations | 1 day (D1) in each treatment period

SECONDARY OUTCOMES:
Measurement of serum insulin concentrations | 1 day (D1) in each treatment period
Measurement of serum C-peptide concentrations | 1 day (D1) in each treatment period
Measurement of plasma glucagon concentrations | 1 day (D1) in each treatment period
Measurement of plasma lixisenatide concentrations | 1 day (D1) in each treatment period
Number of patients with hypoglycemic events | Up to 2 weeks after each treatment
Number of patients with adverse events | Up to 2 weeks after each treatment
Measurement of anti-lixisenatide antibodies | 2 days (prior to first dosing and end of study visit)
Measurement of anti-insulin antibodies | 2 days (prior to first dosing and end of study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 392001, Fukuoka, Japan

REFERENCES:
- [Result] Inoue M, Lorenz M, Muto H, Wesch R, Hashimoto Y. Effect of a single dose of insulin glargine/lixisenatide fixed ratio combination (iGlarLixi) on postprandial glucodynamic response in Japanese patients with type 2 diabetes mellitus: A phase I randomized trial. Diabetes Obes Metab. 2019 Aug;21(8):2001-2005. doi: 10.1111/dom.13757. Epub 2019 May 24. PMID 31050109